CLINICAL TRIAL: NCT05961124
Title: A Phase II, Single-Arm Trial Assessing Alternative Dosing Of Niraparib To Decrease Dose Interruption In First Line Maintenance Treatment For Ovarian Cancer: Dose Escalation
Brief Title: Alternative Dosing Of Niraparib To Decrease Dose Interruption In First Line Maintenance Treatment For Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5397
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-08

CONDITIONS: Ovarian Cancer; Stage III Ovarian Cancer; Stage IV Ovarian Cancer; High Grade Ovarian Serous Adenocarcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm- Niraparib (Experimental): Oral niraparib will be administered in a dose escalation design where patients will start at a dose of 100 mg PO daily for the first two cycles, then 200 mg PO daily for the third and fourth cycle. Patients will remain on the individualized dose until either they experience an adverse event and require a dose reduction or they have disease progression.
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Niraparib (Zejula) will be administered as an oral treatment once daily (continuously in a 28-day cycle). Niraparib will be administered in a dose escalation design where patients will start at a dose of 100 mg PO daily for the first two cycles (28-days each cycle), if tolerated, the dose will be increased to 200 mg PO daily for the third and fourth cycle.
  Other Names: Zejula

SUMMARY:
The goal of this clinical trial is to test alternative dosing of niraparib in patients with newly diagnosed high-grade, advanced stage ovarian cancer. The main questions it aims to answer are:

What is the incidence of hematologic and other adverse events? What is the incidence of dose interruption, dose reduction and discontinuation? What is the length of time of progression-free survival at 24 months?

DETAILED DESCRIPTION:
This is a single arm phase II study in patients with newly diagnosed high-grade, advanced stage ovarian cancer. Patients must have received a minimum of 4 cycles of front-line platinum-based chemotherapy with a complete response or partial response (no measurable lesion >1 cm and normal cancer antigen (CA -25) after completion of chemotherapy) and primary or interval debulking surgery. This study aims to evaluate the incidence of hematologic and other adverse events and the incidence of dose interruption, dose reduction and discontinuation, and progression-free survival at 24 months with a niraparib dose escalation design. Study enrollment is planned to include 40 patients at one site.

ELIGIBILITY:
Inclusion Criteria

1. Patients must be able to understand the study, agree to participate and provide written, informed consent
2. Patients must be female and age >/= 18 years of age
3. Newly diagnosed, histologically confirmed, high-grade serous and grade 3 endometrioid ovarian, primary peritoneal, or fallopian tube cancer undergoing frontline treatment
4. Stage III and IV cancer according to International Federation of Gynecology and Obstetrics (FIGO) 2018 criteria and all patients undergoing neoadjuvant chemotherapy (NACT)
5. Patients must meet the following front-line treatment requirements:

   i. Patients must have completed a minimum of 4 cycles of platinum-based chemotherapy (carboplatin, cisplatin, oxaliplatin). Primary or interval debulking therapy and intraperitoneal chemotherapy are allowed.

   ii. Patients must have a complete response or partial tumor response (no lesion >1cm) to platinum-based regimen

   iii. CA-125 must be either:
   1. CA-125 in normal range or
   2. CA-125 decreased by 90% during front-line treatment and stable for a minimum of 7 days (does not increase by more than 15%) iv. Study drug can start within 12 weeks of completing chemotherapy
6. Patients must be post-menopausal with no menses for >1 year, or surgically sterilized, or willing to use adequate contraception to prevent pregnancy or abstain from intercourse and agrees not to donate eggs for the purpose of reproduction from study enrollment until 6 months following the last dose of treatment.

   i. Patients of childbearing potential must have a negative serum or urine pregnancy test (beta human chorionic gonadotropin [hcg]) within 3 days prior to receiving the first dose of study treatment.
7. Eastern Cooperative Oncology Group (ECOG) status of 0 or 1
8. Patients must have adequate organ function at enrollment, as follows:

   i. Absolute neutrophil count >/= 1.5 x109/L ii. Platelets >/= 100 x109/L iii. Hemoglobin >/= 100 g/L without transfusion iv. Creatinine clearance >/= 60 mL/min using the Cockcroft-Gault equation v. Total bilirubin </= 1.5 times the upper limit of normal (ULN) or direct bilirubin < 1 times the upper limit of normal vi. Aspartate aminotransferase and Alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN
9. Patients with hypertension should have their blood pressure adequately treated and controlled prior to starting study treatment
10. Patients must be able to take oral medications
11. Patients must agree to complete blood samples prior to cycle 1, then weekly for the first month and as outlined in the protocol

Exclusion Criteria:

1. Patient's age is <18 years.
2. Patient who are pregnant, breastfeeding, or expecting to conceive children during the study treatment of for 6 months after completion of the study treatment.
3. Patients with a known hypersensitivity to niraparib or any of its components
4. Patients who have received a poly adenosine diphosphate-ribose polymerase (PARP) inhibitor as part of their previous treatment or participated in a trial where PARP inhibitors were administered in one arm of the trial.
5. Patients enrolled in another investigational trial
6. Patients who received another investigational therapy within 4 weeks or 5 halflives of the investigational agent, whichever is longer
7. Patients with previous persistent (>4 weeks) or >/= grade 3 hematologic toxicity or fatigue from prior cancer therapy.
8. Patients with known history of myelodysplastic syndrome or pre-treatment cytogenetic testing at risk for myelodysplastic syndrome or acute myeloid leukemia
9. Patients receiving concurrent, prohibited medications
10. Patients with previous major surgery within 3 weeks of starting study treatment and must have recovered from any effects of previous surgery.
11. Patients with ascites drained within 4 weeks of starting study treatment
12. Patients receiving palliative radiotherapy to >20% of bone marrow within 2 weeks or any other radiotherapy within 1 week of study treatment
13. Patients receiving a transfusion (platelets or red blood cells) within 4 weeks of treatment
14. Patients planning to donate blood during the study or 90 days after treatment.
15. Patients with a diagnosis of another invasive cancer (other than ovarian cancer), within 2 years prior to randomization (except basal or squamous cell carcinoma of the skin that has been definitively treated i. Patients with uncontrolled brain or leptomeningeal metastases. Controlled brain or leptomeningeal metastasis is defined as: ii. Central nervous system disease that has undergone treatment with radiation or chemotherapy > 1 month before study entry
16. No new or progressive signs or symptoms, stable steroid dose x 4 weeks or not taking steroids
17. Patients considered poor medical risk due to serious, uncontrolled medical disorder, non-malignant systemic disease, or active uncontrolled infection i. Patients with known HIV considered high risk for serious and fatal outcome
18. Patients with evidence of any condition, therapy, or laboratory abnormality that might confound study results or patient participation for full duration of study (Ex. Myelodysplastic syndrome, anemia, leukopenia, neutropenia, thrombocytopenia, etc)
19. Patients who are immunocompromised (Patients with splenectomy are allowed)
20. Patients with known, active hepatic disease (Ex. Hepatitis B or C), active biliary disease (exceptions for Gilbert's syndrome, asymptomatic gallstones, liver metastases or otherwise stable chronic liver disease as per investigator assessment)
21. Patients with QT prolongation >470 milliseconds at screening
22. Patients with a known breast cancer susceptibility gene (BRCA1 and 2) mutation (as they routinely receive olaparib at our institution) If BRCA unknown they are not excluded.
23. Patients with a history of posterior reversible encephalopathy syndrome (PRES)
24. Patients who have had a live vaccine within 30 days of planned start date of study treatment
25. Patients with gastrointestinal abnormalities that may limit absorption
26. Patients with significant cardiovascular disease
27. Patients undergoing serial blood counts to achieve a value to meet eligibility
28. Patients receiving blood product transfusions in order to meet eligibility criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of thrombocytopenia | 2 years
  Incidence of thrombocytopenia <100 x 109/L requiring a treatment interruption

SECONDARY OUTCOMES:
Incidence of dose reduction due to thrombocytopenia | 2 years
Incidence of discontinuation due to thrombocytopenia | 2 years
Incidence of other hematologic toxicity | 2 years
Incidence of dose reduction due to other hematologic toxicity | 2 years
Incidence of discontinuation due to other hematologic toxicity | 2 years
Incidence of other toxicities | 2 years
Incidence of dose reduction due to other toxicities | 2 years
Incidence of discontinuation due to other toxicities | 2 years
Incidence of discontinuation due to disease progression | 2 years
Incidence of discontinuation for other reasons | 2 years
Progression-free survival at 24 months | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Allan Covens, MD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No